CLINICAL TRIAL: NCT07261774
Title: The Impact of Extreme Heat Waves and Air Pollution on the Prognosis of Chronic Airway Diseases
Status: Completed | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Sibel Naycı, Prof. Dr., Mersin University
Other Study IDs: MU-2024/097
Record Dates: First submitted 2025-08-29; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Asthma (Diagnosis); COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Asthma; COPD; Extreme Heatwave; Air Pollution; Climate Change
MeSH Terms: conditions — Asthma; Disease; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma Group: Patients with physician-diagnosed asthma who met the inclusion criteria and were followed during periods of extreme heat waves and normal seasonal weather.
- COPD Group: Patients with physician-diagnosed chronic obstructive pulmonary disease (COPD) who met the inclusion criteria and were followed during periods of extreme heat waves and normal seasonal weather.

SUMMARY:
Extreme heat waves (EHW) and air pollution exacerbate chronic airway diseases, but little is known about how these environmental stressors affect quality of life, airway inflammation, symptom control, and pulmonary function. This study was designed to determine the impact of EHW and air pollution on asthma and COPD.

This was a prospective cohort study conducted among individuals with asthma and COPD in Mersin, Türkiye, between February 14 and December 1, 2024. Meteorological and air quality index (AQI) data were obtained from official sources. Participants underwent pulmonary function tests (PFTs) and fractional exhaled nitric oxide (FeNO) measurements during periods of normal weather conditions and repeated assessments during documented EHW periods. Patient-reported outcomes included the Asthma Control Test (ACT) and Asthma Quality of Life Questionnaire (AQLQ) for asthma, and the Modified Medical Research Council (mMRC) scale and COPD Assessment Test (CAT) for COPD. Exacerbation episodes requiring systemic corticosteroid use or hospitalization were also recorded.

The study aimed to evaluate the effects of EHW and air pollution on disease control, quality of life, lung function, airway inflammation, and exacerbation burden in patients with asthma and COPD.

DETAILED DESCRIPTION:
Climate change has led to a global increase in temperatures, and according to NASA, 2024 was the hottest year on record since 1850. Extreme heatwaves (EHW) represent one of the most significant manifestations of this crisis. While the adverse effects of air pollution on chronic respiratory diseases are well documented, the impact of extreme heatwaves on asthma and chronic obstructive pulmonary disease (COPD) has received less attention.

This study was designed to prospectively evaluate the effects of extreme heatwaves and air pollution on patients with asthma and COPD. The study was conducted in Mersin, Türkiye, between February and December 2024. Individuals with physician-diagnosed asthma or COPD who attended the outpatient clinic were enrolled.

Baseline assessments were performed on days with normal seasonal weather. Lung function was measured using spirometry, and airway inflammation was assessed using fractional exhaled nitric oxide (FeNO). Symptom control and quality of life were measured using validated questionnaires: the Asthma Control Test (ACT) and Asthma Quality of Life Questionnaire (AQLQ) for patients with asthma, and the Modified Medical Research Council (mMRC) scale and COPD Assessment Test (CAT) for patients with COPD.

Meteorological variables, including temperature, humidity, and wind, as well as daily air pollution levels, were obtained from official sources. On documented extreme heatwave days, participants were recalled for follow-up visits. At these visits, spirometry, FeNO, and questionnaire assessments were repeated. Information regarding exacerbation episodes requiring systemic corticosteroid use or hospitalization during the study period was also collected.

The study was designed to compare patient-level outcomes between normal weather days and extreme heatwave days. The overall objective was to investigate how environmental stressors such as heat and air pollution influence disease control, quality of life, symptoms, lung function, and airway inflammation in patients with asthma and COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Provision of written informed consent

For the asthma group:

- Diagnosis of asthma for at least 6 months according to the GINA 2024 guidelines

Variable respiratory symptoms together with documented variable expiratory airflow limitation, demonstrated by at least one of the following:

* Positive bronchodilator reversibility test (>12% and >200 mL increase in FEV1 10-15 minutes after 400 μg salbutamol)
* Peak expiratory flow (PEF) variability (>10% average daily PEF variability over 2 weeks)
* Positive delayed reversibility (improvement in lung function after 4 weeks of anti-inflammatory treatment with >12% and >200 mL increase in FEV1 or >20% increase in PEF)
* Positive bronchial provocation test (≥20% fall in FEV1 with standard doses of methacholine or histamine)
* Stable disease for at least 4 weeks prior to enrollment

For the COPD group:

* Diagnosis of COPD for at least 6 months according to the GOLD 2024 guidelines (post-bronchodilator FEV1/FVC <70% in the presence of compatible clinical findings)
* Stable disease for at least 4 weeks prior to enrollment

Exclusion Criteria:

* Presence of other pulmonary diseases apart from asthma or COPD (e.g., interstitial lung diseases, pleural diseases, pulmonary vascular diseases)
* Pregnant women
* History of cancer within the past 5 years
* Previous lung surgery
* Active pulmonary tuberculosis
* Respiratory tract infection within the last 4 weeks
* Presence of significant extrapulmonary disease that may affect lung function (e.g., cerebrovascular disease, acute myocardial infarction)
* Active smoking within the past year
* Residence outside the central district of Mersin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years) diagnosed with asthma according to the GINA 2024 guidelines or COPD according to the GOLD 2024 guidelines, who are in a stable phase for at least four weeks. Participants must provide written informed consent and reside within the central district of Mersin. Patients with other chronic lung diseases, history of lung surgery, recent respiratory infections, active tuberculosis, significant comorbidities affecting lung function, pregnancy, active smoking within the past year, cancer history within the past five years, or those living outside Mersin city center will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in FeNO levels during extreme heat waves vs seasonal normal conditions | Participants were evaluated twice over a 292-day period, from February 14, 2024, to December 1, 2024 (once during seasonal normal conditions and once during extreme heat waves).
  Fractional exhaled nitric oxide (FeNO) (parts per billion (ppb)) measured using the Bedfont® NObreath device.

SECONDARY OUTCOMES:
Exacerbation frequency in asthma and COPD patients during extreme heat waves vs seasonal normal conditions | Participants were evaluated twice over a 292-day period, from February 14, 2024, to December 1, 2024 (once during seasonal normal conditions and once during extreme heat waves).
  Exacerbations (number of events per participant) defined as events requiring systemic corticosteroid use or hospitalization.

OTHER OUTCOMES:
2. Change in FEV1 during extreme heat waves vs seasonal normal conditions | Participants were evaluated twice over a 292-day period, from February 14, 2024, to December 1, 2024 (once during seasonal normal conditions and once during extreme heat waves).
  FEV1 (liters and % predicted) measured with a hospital-based spirometer.
3. Change in FVC during extreme heat waves vs seasonal normal conditions | Participants were evaluated twice over a 292-day period, from February 14, 2024, to December 1, 2024 (once during seasonal normal conditions and once during extreme heat waves).
  FVC (liters and % predicted) measured with a hospital-based spirometer.
4. Change in ACT score (Asthma Control Test) during extreme heat waves vs seasonal normal conditions | Participants were evaluated twice over a 292-day period, from February 14, 2024, to December 1, 2024 (once during seasonal normal conditions and once during extreme heat waves).
  Description: ACT score (range 5-25, higher scores = better asthma control).
Change in AQLQ score (Asthma Quality of Life Questionnaire) during extreme heat waves vs seasonal normal conditions | Participants were evaluated twice over a 292-day period, from February 14, 2024, to December 1, 2024 (once during seasonal normal conditions and once during extreme heat waves).
  AQLQ score (range 1-7, higher scores = better quality of life).
Change in mMRC score (Modified Medical Research Council Dyspnea Scale) during extreme heat waves vs seasonal normal conditions | Participants were evaluated twice over a 292-day period, from February 14, 2024, to December 1, 2024 (once during seasonal normal conditions and once during extreme heat waves).
  mMRC score (range 0-4, higher scores = worse dyspnea).
Change in CAT score (COPD Assessment Test) during extreme heat waves vs seasonal normal conditions | Participants were evaluated twice over a 292-day period, from February 14, 2024, to December 1, 2024 (once during seasonal normal conditions and once during extreme heat waves).
  CAT score (range 0-40, higher scores = worse quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Faculty of Medicin, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No